CLINICAL TRIAL: NCT05364827
Title: Computed Tomography Coronary Angiography (CTCA) Prior to Chronic Total Occlusion (CTO) Percutaneous Coronary Intervention (PCI) - a Feasibility Study
Brief Title: CT Coronary Angiography Prior to CTO PCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Vinoda Sharma, Consultant Interventional Cardiologist, Sandwell & West Birmingham Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 293244
Record Dates: First submitted 2021-11-04; First posted 2022-05-06 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: computed tomography coronary angiography (CTCA); CTO

STUDY DESIGN:
Intervention Model Description: Prospective randomised feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CTCA prior to CTO PCI (Experimental): A diagnostic CTCA will be conducted prior to CTO PCI by at a level 2 CTCA trained operator. The results will be discussed with the CTO operator prior to the CTO PCI.
  Interventions: Diagnostic Test: CTCA
- No CTCA prior to CTO PCI (No Intervention): Patients will be listed directly for the CTO PCI procedure without undergoing CTCA prior

INTERVENTIONS:
Diagnostic Test: CTCA — CTCA performed in intervention arm patients prior to CTO PCI
  Arms: CTCA prior to CTO PCI

SUMMARY:
A Chronic Total Occlusion or CTO of a coronary artery is a an artery that has been blocked for >/= 3 months. More than a decade ago, patients with such coronary artery blockage would have been sent for Coronary Artery Bypass Graft (CABG) surgery. Newer tools and techniques have facilitated the opening (angioplasty or percutaneous coronary intervention (PCI)) of such occluded arteries- however success is not 100% unlike in simple coronary blockages.

Computed Tomography Coronary Angiography (CTCA) identifies the artery path and characteristics of the CTO including calcification - the latter many times is the reason for failure to cross the CTO.

The investigators aim to conduct a feasibility study to assess the effectiveness of CTCA prior to CTO PCI by randomizing suitable CTO patients to CTCA or direct CTO PCI.

20 patients will be randomized 1:1 using the sealed envelope technique and compared for:

Primary endpoint:

CTO PCI success rate in CTCA arm versus no CTCA arm

Secondary endpoints:

i. Angina by the Seattle Angina Questionnaire (SAQ) at 6 months (range 0-100, lower score worse, higher scores better, based on 5 characteristics - severity, frequency, treatment satisfaction and quality of life scores).

ii. Compare the number of patients who required a second CTO PCI procedure in the CTCA arm versus no CTCA arm iii. Procedural differences between the intervention CTCA arm versus no CTCA arm including: Health Economics: Cost saved per patient due to improved success and reduction in readmission or further procedure CTO PCI efficiency: Wire crossing time, Procedure time CTO PCI safety outcomes: Procedural complications (Ellis perforation, tamponade, acute kidney injury/contrast induced nephropathy, access site bleeding, donor vessel injury), Radiation: CTCA dose, CTO PCI dose, and combined CTCA and CTO PCI dose. Contrast: CTCA volume, CTO PCI volume, and combined CTCA and CTO PCI volume Change in CTO PCI strategy hierarchy as a result of the CTCA review

Patients will have a telephonic follow up at 6 months to assess angina ( by the Seattle Angina Questionnaire)

DETAILED DESCRIPTION:
Computed Tomography Coronary Angiography (CTCA) prior to Chronic Total Occlusion (CTO) Percutaneous Coronary Intervention (PCI) - a feasibility study

Summary of Trial design:

Randomised, prospective, single centre feasibility study of CTCA prior to CTO PCI

Site and Chief Investigator:

Sandwell and West Birmingham NHS Trust, Birmingham, United Kingdom Vinoda Sharma

Participant population Patients undergoing CTO PCI Planned sample size 20 Number of sites 1 Intervention duration Prior to index CTO PCI procedure Follow up duration 6 months Planned trial duration 1 year Primary objective: To determine if CTCA prior to CTO PCI results in improved procedural success rate? Secondary objectives: i) To determine if CTCA prior to CTO PCI results in improved angina as determined by Seattle Angina Questionnaire (SAQ)? ii) To determine if CTCA prior to CTO PCI reduces the need for a second procedure due to improved procedural success rate? iii) Are there procedural differences between the intervention arm (CTCA) and usual care Intervention Randomised to CTCA versus no CTCA prior to CTO PCI

ABBREVIATIONS:

AUC: Area Under the Curve

CABG: Coronary Artery Bypass Graft

CAD: Coronary Artery Disease

CTCA: Computed Tomography Coronary Angiogram

CTO: Chronic Total Occlusion

J-CTO: Japanese Chronic Total Occlusion NHS: National Health Service

PCI: Percutaneous Coronary Intervention

QALYS: Quality Adjusted Life Years

QoL: Quality of Life

SAQ: Seattle Angina Questionnaire

UK: United Kingdom

Trial Protocol Synopsis Item Description

Title Computed Tomography Coronary Angiography (CTCA) prior to Chronic Total Occlusion (CTO) Percutaneous Coronary Intervention (PCI)

Introduction

Description of research question Null Hypothesis:

CTCA performed prior to CTO PCI will not improve procedural success

Existing knowledge:

A chronic total occlusion (CTO) is present in 15-20% of patients with angina who are referred for coronary angiography. Due to the complexity of occlusive coronary artery disease (CAD), including a high prevalence of calcium and tortuosity within long segments of disease, CTO PCI is associated with higher procedural complication rates. Inability to detect the intraluminal path in the CTO artery, combined with calcification and tortuosity can result in unsuccessful guidewire crossing and procedural failure.

Successful CTO PCI has been shown to improve Quality of Life (QoL) at 12 months. These patients are more likely to be angina free at 12 months as assessed by the Seattle Angina Questionnaire (SAQ) (7, 8). CTO PCI in symptomatic patients is cost effective and results in greater quality-adjusted-life-years (QALYS).

CTO percutaneous coronary intervention (PCI) procedure success rates increased from 68% to 79% between 2000 and 2011, and are as high as 90% when performed by high-volume CTO operators (2, 3). Complexity of the CTO is determined by several factors and several CTO complexity scores, derived from (invasive) angiographic lesion and clinical characteristics, have been shown to correlate with procedural success and complication rates (JCTO, PROGRESS, RECHARGE, Euro-CASTLE).

The most commonly utilized score is the J-CTO (Multicenter Chronic Total Occlusion Registry of Japan) which assigns a score of 1 each to the angiographic CTO proximal cap (tapered or blunt), calcification, tortuosity (>45degrees), lesion length (≥20mm) and previous failure, with a maximum score =5. Scores ≥2 are considered CTOs that are difficult to perform and require advanced techniques for successful revascularization.

In a proportion of these patients, the first procedure either fails completely or partially succeeds in forming a tract within the occluded artery but this is inadequate for stent delivery and the patient requires a second procedure, occasionally a third for complete success and reconstruction of the fully occluded artery.

Angiographically, the CTO artery usually shows a short proximal portion of dye filled artery prior to the occlusion. In most patients there are some collaterals from the contralateral coronary artery which try to fill part of the occluded CTO artery. However the actual body of the CTO is not visible angiographically.

Computed Tomography Coronary Angiography (CTCA) can delineate the coronary anatomy in 3-dimensions, determining atherosclerotic plaque and occlusion location, severity and morphology. This makes it an attractive modality to assess the coronary CTO. Development of a CTCA based complexity score for stratifying CTOs by difficulty resulted in the CT-RECTOR score (Computed Tomography Registry of Chronic Total Occlusion Revascularization, table 1). Variables included in this score are multiple occlusions, blunt stump, severe calcification, bending, duration of CTO ≥12 months and previously failed PCI (all scored 1). The CT-RECTOR score correlates with the J-CTO score and has a better area under ROC curve (ROC AUC 0.83 for CT-RECTOR score and 0.71 for J-CTO, p < 0.001) and predicts CTO PCI success.

The role of routine CTCA pre-CTO PCI is as yet undefined as current practice involves the use of CTCA in patients who have had an unsuccessful CTO PCI attempt or previous coronary artery bypass grafting (CABG).

Need for a feasibility study:

Current practice at our center involves the use of CTCA in patients who have had an unsuccessful CTO PCI attempt or previous coronary artery bypass grafting (CABG) but the role of routine CTCA pre-CTO PCI is as yet undefined.

The small additional investment of a CTCA could help plan/improve a complex procedure and may reduce the need for additional procedures and readmissions.

The mean acute treatment cost of a CTO PCI is approximately (combined day-case -ordinary elective spell) £6933 whereas the approximate cost of a CTCA is £360 (as per local billing). Elective readmission for a failed CTO PCI procedure would entail an additional financial (to the provider) and emotional cost (to the patient).

The cost of an additional CTO PCI procedure aside, readmission and bed charges themselves can reach £1000/day (readmission =£255/day) and bed cost=£600/day). Including the cost of a second CTO PCI procedure (combined day-case -ordinary elective spell) £6933 - the overall cost can total to £10,000. In contrast, the cost of a CTCA is £360 (as per local billing).

Financial costs are one part of the issue, but a second CTO PCI procedure can also heighten patient anxiety and discomfort which are well known in patients prior to any PCI.

A feasibility study will help establish the role of a CTCA prior to CTO PCI to positively influence strategy and/or outcomes.

Methods:

Study setting: Sandwell and West Birmingham NHS Trust, Birmingham, United Kingdom.

Trial design: This is a randomized (1:1), prospective, single center study. Patients with suitable eligibility criteria will be included and randomized to CTCA or no CTCA prior to CTO PCI and the primary and secondary outcomes compared between the two groups

Sample size: This is a feasibility study- to ensure completion within a year, the investigators have estimated 20 patients, randomized 1:1 to each arm (10 patients per arm) as a sample size in a moderate size hospital which performs approximately 100 CTO PCIs annually.

Intervention assignment: Block randomization with sealed envelope technique.

Participant/project timeline: To complete: 1 year

Data collection, management and analysis

* eCRF (electronic Case Report Form) and online database to collect demographic, procedural and SAQ information
* SAQ at 6 months post PCI
* Blood samples pre and post PCI
* Comparison of demographics, procedural details, procedural success and complications, bloods, SAQ, and financial cost between the CTCA and non-CTCA groups
* Categorical variables will be presented as percentage and compared with the chi square or Fisher's test
* Continuous variables will be presented as median (range) and compared with student's t-test or Mann Whitney test.
* In addition, modelling will be performed by binary logistic regression analysis to predictors of CTO PCI success.

Monitoring: CTO PCI procedural adverse events will be reported as usual on the national database and this data will be collected in the eCRF.

Ethics: Ethical approval for this prospective study has been obtained All patients will be consented prior to inclusion in this study.

Blood: Routine blood tests will be performed immediately before the CTO PCI and after the procedure prior to discharge-this is standard of care.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* CTO with J-CTO score≥2
* Appropriate indication for CTO PCI
* Adequate CTCA images for analysis

Exclusion Criteria:

* <18 years of age
* CTO with J-CTO score<2
* Inadequate/degraded CTCA images
* Pregnant/lactating women
* Patients with severe contrast allergy
* Patients unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 24 hours = Day 0 of the index CTO PCI procedure
  CTO PCI success rate in CTCA arm versus no CTCA arm

SECONDARY OUTCOMES:
i. Angina | 6 months
  i. Angina by the SAQ score
ii. More than one CTO PCI procedure required | 24 hours = Day 0 of the index CTO PCI procedure
  ii. Compare the number of patients who required a second CTO PCI procedure in the CTCA arm versus no CTCA arm
iii. Procedural differences between the intervention CTCA arm versus no CTCA arm-health economics | One year = At the end of the study
  Cost saved per patient based on success and reduction in repeat procedure and readmission
iv. Procedural differences between the intervention CTCA arm versus no CTCA arm-CTO PCI wire crossing time | 24 hours = Day 0 of the index CTO PCI procedure
  Time taken to cross the CTO in minutes
v. Procedural differences between the intervention CTCA arm versus no CTCA arm-CTO PCI total procedure time | 24 hours = Day 0 of the index CTO PCI procedure
  Time taken to complete the CTO PCI procedure in minutes
vi. CTO PCI safety outcomes: Procedural complications (Ellis perforation, tamponade, acute kidney injury/contrast induced nephropathy, access site bleeding, donor vessel injury) | 24 hours = Day 0 of the index CTO PCI procedure except acute kidney injury which will be based on blood tests 48 hours after completion of the procedure
  Any complication that is procedure related
vii. CTO PCI safety outcomes: Radiation: CTCA dose, CTO PCI dose, and combined CTCA and CTO PCI dose | 24 hours = Day 0 of the index CTO PCI procedure
  Total radiation dose at the end of the procedure and additive in the CTCA arm versus the no CTCA arm
viii. CTO PCI safety outcomes: Contrast: CTCA volume, CTO PCI volume, and combined CTCA and CTO PCI volume | 24 hours = Day 0 of the index CTO PCI procedure
  Total contrast dose in milliliters at the end of the procedure and additive in the CTCA arm versus the no CTCA arm
ix. Change in CTO PCI strategy hierarchy as a result of the CTCA review : Initial procedure strategy in planning versus actual initial and final procedure strategy | 24 hours = Day 0 of the index CTO PCI procedure
  Any change in the CTO PCI strategy due to CTCA

CONTACTS AND LOCATIONS:
Locations (1):
- SWBH NHS Trust, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Result] Walsh SJ, Hanratty CG, McEntegart M, Strange JW, Rigger J, Henriksen PA, Smith EJ, Wilson SJ, Hill JM, Mehmedbegovic Z, Chevalier B, Morice MC, Spratt JC. Intravascular Healing Is Not Affected by Approaches in Contemporary CTO PCI: The CONSISTENT CTO Study. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1448-1457. doi: 10.1016/j.jcin.2020.03.032. PMID 32553333
- [Result] Tajti P, Brilakis ES. Chronic Total Occlusion Percutaneous Coronary Intervention: Evidence and Controversies. J Am Heart Assoc. 2018 Jan 12;7(2):e006732. doi: 10.1161/JAHA.117.006732. No abstract available. PMID 29330258
- [Result] Werner GS, Martin-Yuste V, Hildick-Smith D, Boudou N, Sianos G, Gelev V, Rumoroso JR, Erglis A, Christiansen EH, Escaned J, di Mario C, Hovasse T, Teruel L, Bufe A, Lauer B, Bogaerts K, Goicolea J, Spratt JC, Gershlick AH, Galassi AR, Louvard Y; EUROCTO trial investigators. A randomized multicentre trial to compare revascularization with optimal medical therapy for the treatment of chronic total coronary occlusions. Eur Heart J. 2018 Jul 7;39(26):2484-2493. doi: 10.1093/eurheartj/ehy220. PMID 29722796
- [Result] Chan PS, Jones PG, Arnold SA, Spertus JA. Development and validation of a short version of the Seattle angina questionnaire. Circ Cardiovasc Qual Outcomes. 2014 Sep;7(5):640-7. doi: 10.1161/CIRCOUTCOMES.114.000967. Epub 2014 Sep 2. PMID 25185249
- [Result] Spertus JA, Winder JA, Dewhurst TA, Deyo RA, Prodzinski J, McDonell M, Fihn SD. Development and evaluation of the Seattle Angina Questionnaire: a new functional status measure for coronary artery disease. J Am Coll Cardiol. 1995 Feb;25(2):333-41. doi: 10.1016/0735-1097(94)00397-9. PMID 7829785
- [Result] Gada H, Whitlow PL, Marwick TH. Establishing the cost-effectiveness of percutaneous coronary intervention for chronic total occlusion in stable angina: a decision-analytic model. Heart. 2012 Dec;98(24):1790-7. doi: 10.1136/heartjnl-2012-302581. Epub 2012 Oct 4. PMID 23038791
- [Result] Grantham JA, Jones PG, Cannon L, Spertus JA. Quantifying the early health status benefits of successful chronic total occlusion recanalization: Results from the FlowCardia's Approach to Chronic Total Occlusion Recanalization (FACTOR) Trial. Circ Cardiovasc Qual Outcomes. 2010 May;3(3):284-90. doi: 10.1161/CIRCOUTCOMES.108.825760. Epub 2010 Apr 13. PMID 20388873
- [Result] Patel VG, Brayton KM, Tamayo A, Mogabgab O, Michael TT, Lo N, Alomar M, Shorrock D, Cipher D, Abdullah S, Banerjee S, Brilakis ES. Angiographic success and procedural complications in patients undergoing percutaneous coronary chronic total occlusion interventions: a weighted meta-analysis of 18,061 patients from 65 studies. JACC Cardiovasc Interv. 2013 Feb;6(2):128-36. doi: 10.1016/j.jcin.2012.10.011. Epub 2013 Jan 23. PMID 23352817
- [Result] Sharma V, Jadhav ST, Harcombe AA, Kelly PA, Mozid A, Bagnall A, Richardson J, Egred M, McEntegart M, Shaukat A, Oldroyd K, Vishwanathan G, Rana O, Talwar S, McPherson M, Strange JW, Hanratty CG, Walsh SJ, Spratt JC, Smith WH. Impact of proctoring on success rates for percutaneous revascularisation of coronary chronic total occlusions. Open Heart. 2015 Mar 28;2(1):e000228. doi: 10.1136/openhrt-2014-000228. eCollection 2015. PMID 25852949
- [Result] Morino Y, Abe M, Morimoto T, Kimura T, Hayashi Y, Muramatsu T, Ochiai M, Noguchi Y, Kato K, Shibata Y, Hiasa Y, Doi O, Yamashita T, Hinohara T, Tanaka H, Mitsudo K; J-CTO Registry Investigators. Predicting successful guidewire crossing through chronic total occlusion of native coronary lesions within 30 minutes: the J-CTO (Multicenter CTO Registry in Japan) score as a difficulty grading and time assessment tool. JACC Cardiovasc Interv. 2011 Feb;4(2):213-21. doi: 10.1016/j.jcin.2010.09.024. PMID 21349461
- [Result] Christopoulos G, Kandzari DE, Yeh RW, Jaffer FA, Karmpaliotis D, Wyman MR, Alaswad K, Lombardi W, Grantham JA, Moses J, Christakopoulos G, Tarar MNJ, Rangan BV, Lembo N, Garcia S, Cipher D, Thompson CA, Banerjee S, Brilakis ES. Development and Validation of a Novel Scoring System for Predicting Technical Success of Chronic Total Occlusion Percutaneous Coronary Interventions: The PROGRESS CTO (Prospective Global Registry for the Study of Chronic Total Occlusion Intervention) Score. JACC Cardiovasc Interv. 2016 Jan 11;9(1):1-9. doi: 10.1016/j.jcin.2015.09.022. PMID 26762904
- [Result] Maeremans J, Spratt JC, Knaapen P, Walsh S, Agostoni P, Wilson W, Avran A, Faurie B, Bressollette E, Kayaert P, Bagnall AJ, Smith D, McEntegart MB, Smith WHT, Kelly P, Irving J, Smith EJ, Strange JW, Dens J. Towards a contemporary, comprehensive scoring system for determining technical outcomes of hybrid percutaneous chronic total occlusion treatment: The RECHARGE score. Catheter Cardiovasc Interv. 2018 Feb 1;91(2):192-202. doi: 10.1002/ccd.27092. Epub 2017 May 4. PMID 28471074
- [Result] Szijgyarto Z, Rampat R, Werner GS, Ho C, Reifart N, Lefevre T, Louvard Y, Avran A, Kambis M, Buettner HJ, Di Mario C, Gershlick A, Escaned J, Sianos G, Galassi A, Garbo R, Goktekin O, Meyer-Gessner M, Lauer B, Elhadad S, Bufe A, Boudou N, Sievert H, Martin-Yuste V, Thuesen L, Erglis A, Christiansen E, Spratt J, Bryniarski L, Clayton T, Hildick-Smith D. Derivation and Validation of a Chronic Total Coronary Occlusion Intervention Procedural Success Score From the 20,000-Patient EuroCTO Registry: The EuroCTO (CASTLE) Score. JACC Cardiovasc Interv. 2019 Feb 25;12(4):335-342. doi: 10.1016/j.jcin.2018.11.020. Epub 2019 Jan 30. PMID 30711551
- [Result] Opolski MP, Achenbach S, Schuhback A, Rolf A, Mollmann H, Nef H, Rixe J, Renker M, Witkowski A, Kepka C, Walther C, Schlundt C, Debski A, Jakubczyk M, Hamm CW. Coronary computed tomographic prediction rule for time-efficient guidewire crossing through chronic total occlusion: insights from the CT-RECTOR multicenter registry (Computed Tomography Registry of Chronic Total Occlusion Revascularization). JACC Cardiovasc Interv. 2015 Feb;8(2):257-267. doi: 10.1016/j.jcin.2014.07.031. PMID 25700748
- See also: Cost of CTO and CTCA in UK, reference #16 — http://improvement.nhs.uk/documents/4980/1920_National_Tariff_Payment_System.pdf

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT05364827/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT05364827/ICF_001.pdf